CLINICAL TRIAL: NCT06435065
Title: Histological and Radiographic Evaluation of the Effects of Direct Pulp Capping Agent on Human Pulp Tissue
Brief Title: Direct Pulp Capping Agent on Human Pulp Tissue
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: DR SURINDER SACHDEVA (Other)
Responsible Party: Sponsor-Investigator, DR SURINDER SACHDEVA, periodontist, Maharishi Markendeswar University (Deemed to be University)
Organization: Maharishi Markendeswar University (Deemed to be University) (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2264
Record Dates: First submitted 2024-05-17; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Reversible Pulpitis
Keywords: DIRCT PULP CAPPING; Biodentine; MTA; TheraCal LC; Tristrontium Aluminate
MeSH Terms: interventions — tricalcium silicate; TheraCal; Pemetrexed

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BIODENTINE (Sham Comparator): DIRECT PULP CAPPING WILL BE DONE USING BIODENTINE AS DIRECT PULP CAPPING AGENT
  Interventions: Drug: Biodentine
- MINERAL TRIOXIDE AGGREGATE (Sham Comparator): DIRECT PULP CAPPING WILL BE DONE USING MTA AS DIRECT PULP CAPPING AGENT
  Interventions: Drug: Mineral Tri-Oxide Aggregate
- THERACAL LC (Sham Comparator): DIRECT PULP CAPPING WILL BE DONE USING THERACAL LC AS DIRECT PULP CAPPING AGENT
  Interventions: Drug: THERACAL LC
- TRISTRONTIUM ALUMINATE (Active Comparator): DIRECT PULP CAPPING WILL BE DONE USING TRISTRONTIUM ALUMINATE AS DIRECT PULP CAPPING AGENT
  Interventions: Drug: TRISTRONTIUM ALUMINATE

INTERVENTIONS:
Drug: Biodentine — DIRECT PULP CAPPINGWILL BE DONE USING BIODENTINE
  Arms: BIODENTINE
Drug: Mineral Tri-Oxide Aggregate — DIRECT PULP CAPPINGWILL BE DONE USING MTA
  Other Names: MTA
  Arms: MINERAL TRIOXIDE AGGREGATE
Drug: THERACAL LC — DIRECT PULP CAPPINGWILL BE DONE USING THERACAL LC
  Arms: THERACAL LC
Drug: TRISTRONTIUM ALUMINATE — DIRECT PULP CAPPINGWILL BE DONE USING TRISTRONTIUM ALUMINATE
  Arms: TRISTRONTIUM ALUMINATE

SUMMARY:
This in- vivo study was conducted to evaluate the response of human pulp tissue following direct pulp capping using four different pulp capping agents in premolars scheduled for extraction in patients undergoing orthodontic treatment.

DETAILED DESCRIPTION:
For the study 40 premolars from patients in the age group of 15-25 years, undergoing orthodontic treatment, in the Department of Orthodontics, MMCDSR, Mullana, Ambala, who had to get their premolars extracted as per their orthodontic treatment plan will be selected.

Only healthy premolars, with no caries, showing no signs and symptoms of pulpitis or periodontal diseases were selected. Medically compromised patients, or teeth with radiographic findings of external/internal resorption, bone loss, or calcifications in the pulp chamber will be excluded from the study. The selected premolars were then randomly divided into four equal groups namely: GROUP I - Direct pulp capping procedure performed using Biodentine. GROUP II - Direct pulp capping procedure performed using MTA. GROUP III - Direct pulp capping procedure performed using TheraCal LC. GROUP IV - Direct pulp capping procedure performed using Tristrontium aluminate.

The direct pulp capping procedure was carried out under rubber dam. The study protocol included class I cavity preparations on the premolars, followed by iatrogenic exposure of the pulp (0.5mm) using a sterile round bur, placement of the direct pulp capping agent according to the material of allotted to the study group. The teeth were permanently restored on the same visit, except for MTA group were the teeth were temporarily restored using Cavit G, and recalled after 1 day for permanent restoration. The patients were then enquired for any 94 SUMMARY 95 symptoms at 1 day and 7 days post operatively. The teeth were then, atraumatically extracted 3 months after the procedure. The extracted teeth were then put to CBCT as well as histopathological examination. Through CBCT evaluation, the completeness of the dentine bridge was evaluated. Histopathological examination was done to examine the pulpal response and the quality of the dentine bridge formed

ELIGIBILITY:
INCLUSION CRITERIA:

* CARIES-free, undamaged mature maxillary and mandibular premolars that were planned for extraction for orthodontic reasons.
* Teeth that show no reaction to percussion.
* Teeth with no previous restorations.
* Teeth that show vitality, when checked with an electric pulp tester.
* Teeth that show no signs of caries or periapical pathology when examined
* radiographically.
* Fully erupted teeth, that allowed proper application of rubber dam.

EXCLUSION CRITERIA:

* caries are present
* Teeth with signs and symptoms of irreversible pulpitis, such as nighttime severe pain
* or spontaneous pain.
* Teeth that show sensitivity to hot and/or cold.
* Radiographic examination reveals any signs of caries, periapical pathology,
* internal/external root resorption, furcal radiolucency/ inter-radicular bone destruction
* and/or calcifications in the pulp chamber or canals.
* Medically compromised patient.
* Pregnant patient.

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
RADIOGRAPHIC EVALUATION OF FOUR DIRECT PULP CAPPING MATERIALS ON HUMAN PULP TISSUE | 90 DAYS
  radiographic examination will be done after 90 days and presence or absence of secondary dentin formation and completeness of the dentinal bride formed will be evaluated by CBCT
HISTOLOGICAL EVALUATION OF FOUR DIRECT PULP CAPPING MATERIALS ON HUMAN PULP TISSUE | 90 DAYS
  Histological examination of the extracted teeth will be done after 90 days and evidence of dentinal bridge formation will be evaluated microscopically

CONTACTS AND LOCATIONS:
Overall Officials: surinder sachdeva, mds, Study Director — professor
Locations (1):
- Swati, Ambāla, Haryana, India

REFERENCES:
- [Background] Parolia A, Kundabala M, Rao NN, Acharya SR, Agrawal P, Mohan M, Thomas M. A comparative histological analysis of human pulp following direct pulp capping with Propolis, mineral trioxide aggregate and Dycal. Aust Dent J. 2010 Mar;55(1):59-64. doi: 10.1111/j.1834-7819.2009.01179.x. PMID 20415913
- [Background] Nowicka A, Lipski M, Parafiniuk M, Sporniak-Tutak K, Lichota D, Kosierkiewicz A, Kaczmarek W, Buczkowska-Radlinska J. Response of human dental pulp capped with biodentine and mineral trioxide aggregate. J Endod. 2013 Jun;39(6):743-7. doi: 10.1016/j.joen.2013.01.005. Epub 2013 Apr 10. PMID 23683272